CLINICAL TRIAL: NCT04281511
Title: A Longitudinal, Observational Biomarker Study in Pancreatic Cancer Patients Receiving Chemotherapy
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Sang Myung Woo, Chief, Senior Scientist, National Cancer Center, Korea
Other Study IDs: NCC2019-0034
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Biomarker; chemotherapy; pharmacogenomic; clinical trials
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — cancer tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Based on the literature, the pancreatic cancer treatment predictor biomarker, which is used in the domestic clinical field, is actually applied to the pancreatic cancer patient cohort of the National Cancer Center.
2. To systematically prospectively identify prospective treatment response biomarkers for Pancreatic Cancer Cohort in the National Cancer Center

DETAILED DESCRIPTION:
1. Immunohistochemistry and gene test for hENT1, DCK, SMAD4, CES2, BRCA 1/2,PALB2, MMRd, MSI, Tumor Ag and etc. on Cancer sample
2. Collect data of Biomarker for pancreatic cancer
3. Compare with Big data and Cohort study in National cancer center
4. The number of subjects is changed by statistical consideration. 218->238

ELIGIBILITY:
Inclusion Criteria:

* Pathologically Confirmed Pancreatic Cancer Patients

Exclusion Criteria:

* Subjects who do not agree with the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pancreatic Cancer Patients
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
median survival | 5 years
  The length of time from either the date of diagnosis or the start of treatment for a disease,the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse
progressive-free survival | 5 years
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse

CONTACTS AND LOCATIONS:
Overall Officials: Sangmyung Woo, Principal Investigator — National Cancer Center
Locations (1):
- NATIONAL CANCER CENTER 323, Ilsan-ro, Ilsandong-gu,, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Result] Farrell JJ, Elsaleh H, Garcia M, Lai R, Ammar A, Regine WF, Abrams R, Benson AB, Macdonald J, Cass CE, Dicker AP, Mackey JR. Human equilibrative nucleoside transporter 1 levels predict response to gemcitabine in patients with pancreatic cancer. Gastroenterology. 2009 Jan;136(1):187-95. doi: 10.1053/j.gastro.2008.09.067. Epub 2008 Oct 7. PMID 18992248
- [Result] Greenhalf W, Ghaneh P, Neoptolemos JP, Palmer DH, Cox TF, Lamb RF, Garner E, Campbell F, Mackey JR, Costello E, Moore MJ, Valle JW, McDonald AC, Carter R, Tebbutt NC, Goldstein D, Shannon J, Dervenis C, Glimelius B, Deakin M, Charnley RM, Lacaine F, Scarfe AG, Middleton MR, Anthoney A, Halloran CM, Mayerle J, Olah A, Jackson R, Rawcliffe CL, Scarpa A, Bassi C, Buchler MW; European Study Group for Pancreatic Cancer. Pancreatic cancer hENT1 expression and survival from gemcitabine in patients from the ESPAC-3 trial. J Natl Cancer Inst. 2014 Jan;106(1):djt347. doi: 10.1093/jnci/djt347. Epub 2013 Dec 3. PMID 24301456
- [Result] Yamada R, Mizuno S, Uchida K, Yoneda M, Kanayama K, Inoue H, Murata Y, Kuriyama N, Kishiwada M, Usui M, Ii N, Tsuboi J, Tano S, Hamada Y, Tanaka K, Horiki N, Ogura T, Shiraishi T, Takei Y, Katayama N, Isaji S. Human Equilibrative Nucleoside Transporter 1 Expression in Endoscopic Ultrasonography-Guided Fine-Needle Aspiration Biopsy Samples Is a Strong Predictor of Clinical Response and Survival in the Patients With Pancreatic Ductal Adenocarcinoma Undergoing Gemcitabine-Based Chemoradiotherapy. Pancreas. 2016 May-Jun;45(5):761-71. doi: 10.1097/MPA.0000000000000597. PMID 26784908
- [Result] Sebastiani V, Ricci F, Rubio-Viqueira B, Kulesza P, Yeo CJ, Hidalgo M, Klein A, Laheru D, Iacobuzio-Donahue CA. Immunohistochemical and genetic evaluation of deoxycytidine kinase in pancreatic cancer: relationship to molecular mechanisms of gemcitabine resistance and survival. Clin Cancer Res. 2006 Apr 15;12(8):2492-7. doi: 10.1158/1078-0432.CCR-05-2655. PMID 16638857
- [Result] Capello M, Lee M, Wang H, Babel I, Katz MH, Fleming JB, Maitra A, Wang H, Tian W, Taguchi A, Hanash SM. Carboxylesterase 2 as a Determinant of Response to Irinotecan and Neoadjuvant FOLFIRINOX Therapy in Pancreatic Ductal Adenocarcinoma. J Natl Cancer Inst. 2015 May 29;107(8):djv132. doi: 10.1093/jnci/djv132. Print 2015 Aug. PMID 26025324